CLINICAL TRIAL: NCT00988546
Title: Evaluation of Computerized Template Entry for C&P Examinations
Brief Title: Evaluation of Computerized Template Entry for Compensation and Pension (C&P) Examinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Speroff, Theodore - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CSRD-000-00F
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Joint Diseases
Keywords: Disability Evaluation; Joint Diseases; Joint Disability
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): exam documentation performed using dictation
  Interventions: Other: Dictation for exam documentation
- 2 (Experimental): exam documentation performed using computer based template
  Interventions: Other: Computer based template for exam documentation

INTERVENTIONS:
Other: Computer based template for exam documentation — exam documentation performed using computer based template
  Arms: 2
Other: Dictation for exam documentation — exam documentation performed using dictation, the standard practice
  Arms: 1

SUMMARY:
The purpose of this study is to compare C&P examination reports performed using a Compensation and Pension Examination Program (CPEP) computerized, templated documentation tool to a customary examination performed and then report dictated in quality, completeness, timeliness and veteran satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for the current study included veterans scheduled for C&P examination of two or fewer joints at VA TVHS.
* No ethnic or racial group or gender was excluded.

Exclusion Criteria:

* Veterans were excluded if they were scheduled:

  1. for examination of more than two joints,
  2. with other requested exam protocols in addition to joints

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-05; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
disability exam report quality | upon completion of report, generally within 3 months

SECONDARY OUTCOMES:
disability exam report data entry time | upon creation of report
disability exam encounter time | upon creation of report
disability exam patient satisfaction | following exam

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Speroff, PhD MS PhD, Principal Investigator — VA Medical Center
Locations (1):
- VA Medical Center, Nashville, Tennessee, United States